CLINICAL TRIAL: NCT05837637
Title: Validation of the Utility of the Vietnamese Smell Identification Test in Vietnamese Patients With Parkinson's Disease
Brief Title: The Vietnamese Smell Identification Test in the Diagnosis of Parkinson's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Center Ho Chi Minh City (UMC) (Other)
Responsible Party: Sponsor
Other Study IDs: 688/HĐĐĐ-ĐHYD
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-04

CONDITIONS: Hyposmia; Parkinson Disease
MeSH Terms: conditions — Anosmia; Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkinson's disease patients: Parkinson's disease patients attend the Parkinson and Movement disorder clinic at Ho Chi Minh University Medical Center
  Interventions: Diagnostic Test: The Vietnamese Smell Identification test (VSIT), the Brief Smell Identification test (BSIT)
- healthy control: The participants including hospital staffs and relatives of patients that matched age and gender
  Interventions: Diagnostic Test: The Vietnamese Smell Identification test (VSIT), the Brief Smell Identification test (BSIT)

INTERVENTIONS:
Diagnostic Test: The Vietnamese Smell Identification test (VSIT), the Brief Smell Identification test (BSIT) — * The VSIT: Odorants used in the VSIT are odorous liquids commercially available in Vietnam. Cotton buds are dipped in diluted odor solution and are used as test materials. The cotton swab is then packaged in a sterile and non-volatile sachet. Participants tore the cotton swab-containing sachet in the direction of the arrow to reveal the bud of the cotton swab and place it approximately 2 cm from the nostrils for 2-3 seconds. The score based on the number of correct answers ranges from 0 to 12.
  * The BSIT: BSIT will be purchased from Sensoics, Inc. and used according to the manufacturer's instructions. Odorants are microencapsulated on the paper and odors are released when the subject uses a pencil to scratch the microcapsule coating. Odorants are placed 2 cm from the both nostrils and participants selected the smell from the answer card containing four options for each odorant. The score based on the number of correct answers ranges from 0 to 12

SUMMARY:
The goal of this observational study is to assess the value of the Vietnamese smell identification test (VSIT) in the diagnosis of Parkinson's disease, and compare it with the commonly used test in the world, Brisk smell identification test (BSIT)

The main questions it aims to answer are:

* The sensitivity, specificity, positive predictive value, and negative predictive value of the VSIT in the diagnosis of Parkinson's disease?
* The sensitivity, specificity, positive predictive value, and negative predictive value of the BSIT in the diagnosis of Parkinson's disease?
* Factors that associated with olfactory identification ability in PD patients?

Process:

* Participants will be assessed cognitive station using MMSE
* Information on socio-demographic including age, gender, education, occupation, place of residence of both groups, and disease-related characteristics will be collected.
* Participants with Parkinson disease will be then assessed with the following instruments: Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS), Hoehn & Yarh scale, and Beck Depression Inventory
* The case and control groups will be assessed by the Vietnamese Smell Identification Test and Brisk Smell Identification Test

DETAILED DESCRIPTION:
Rational Parkinson's disease is one of the most commonly neurodegenerative disorders neurological outbreaks with an incidence in Vietnam of 80-90/100,000 people. It comprises of motor and non-motor symptoms (NMS). Motor symptoms include tremor, bradykinesia, rigidity, gait difficulties, postural instability and falls. Non-motor symptoms are diverse including a wide range of symptoms involving almost systems of the body. A number of nonmotor symptoms may precede motor symptoms by several years, including olfactory dysfunction, constipation, REM sleep behavior disorder, and depression. Since1975, after Ansari and Johnson reported impaired olfactory function in Parkinson's patients, many studies have been conducted with the goal of demonstrating a diminished sense of smell in Parkinson's patients. Recent studies have noted that 70-90% of Parkinson's patients have hyposmia. Current evidence suggests that Parkinson's patients may experience disturbances in various aspects of olfactory function including odor detection, odor discrimination, and odor perception. However, some studies indicated that odor recognition function was more often affected than odor discrimination function. Nowadays, hyposmia is one of the supportive criteria in the diagnosis of Parkinson's disease based on the Parkinson's disease diagnostic criteria of the Movement Disorders Association. Besides, hyposmia when combined with other signs on DAT-Scan and on transcranial Doppler ultrasound help increase the accuracy in diagnosing Parkinson's disease.

There are many different tests available on the market to assess olfactory function for Parkinson's patients, of which the most commonly used tests are UPSIT (University of Pennsylvania Smell Identification Test), B-SIT (Brief Smell Identification test). Identification Test) and Sniffin's Sticks. UPSIT is an odor identification test, developed in 1984 with 40 different odorants. UPSIT has been shown to be highly reliable and valuable in the assessment of odor disorders 19. However, evaluating UPSIT took a long time, so a simpler version of UPSIT with 12 different flavors suitable for many cultures was created called B-SIT. These 12 scents were selected from surveys conducted in several countries in North America, South America, Europe and Asia. In Asia, surveys were conducted in Japan and China. Many studies have shown that B-SIT has good sensitivity and specificity in the diagnosis of Parkinson's disease. However, the popular assessment methods including UPSIT, B-SIT and Sniffin's Sticks were all developed in other parts of the world, so there are many odors in these tests that are not familiar to Vietnamese people. The 12-item Vietnamese smell identification test (VSIT) has been developed to evaluate olfactory function for the Vietnamese population. The VSIT demonstrated good validity and reliability. To date, there have been no studies evaluating the effectiveness of odor identification tests in diagnosing Parkinson's disease in Vietnam. Therefore, investigators conducted this study with the aim to assess the value of the VSIT in the diagnosis of Parkinson's disease, and compare it with the commonly used test in the world, B-SIT.

Primary research objective:

• To determine the sensitivity, specificity, positive predictive value, and negative predictive value of the VSIT in the diagnosis of Parkinson's disease?

Secondary research objective:

* To determine the sensitivity, specificity, positive predictive value, and negative predictive value of the BSIT in the diagnosis of Parkinson's disease?
* To find factors that associated with olfactory identification ability in PD patients?

Approach to participants:

• Patients and controls attending the Parkinson and Movement disorder clinic at UMC will be approached by one of the researchers about the study when the patients come for their regular visit

Research Process:

* Participants will be assessed cognitive station using MMSE
* Information on socio-demographic including age, sex, education, occupation, place of residence of both groups, and disease-related characteristics will be collected.
* Participants with PD will be then assessed with the following instruments: Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS), Hoehn & Yarh scale, and Beck Depression Inventory
* The case and control groups will be assessed by the Vietnamese Smell Identification Test and Brisk Smell Identification Test

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older
* MMSE score > 24
* Clinical diagnosis of Parkinson's disease (for patient group)

Exclusion Criteria:

* History of trauma to the head, history of nasal bone fracture, and history of nasal cosmetic surgery
* Brain neoplasms
* History of stroke, epilepsy
* Secondary Parkinson's and Parkinson's Plus
* Other neurodegenerative diseases, such as Alzheimer's
* Mental disorders, such as schizophrenia, depression
* Upper respiratory tract infections in the 2 weeks
* Pregnancy
* Exposure to medications relating to olfactory reduction, for instance, some particular antibiotics, antiepileptics, antithyroid or benzodiazepines
* Having reported COVID-19 compatible smell symptomatology

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population: Parkinson's disease patients and healthy control
  Target Population:
  1. Parkinson's disease patients attend the Parkinson and Movement disorder clinic at Ho Chi Minh University Medical Center
  Control Population:
  1. The participants included hospital staffs and relatives of patients that matched age and sex
Sampling Method: Non-Probability Sample
Enrollment: 218 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
The VSIT score of both groups | From May 2023 to May 2025
  The VSIT score of both groups will be calculated after testing

SECONDARY OUTCOMES:
The BSIT score of both groups | From May 2023 to May 2025
  The BSIT score of both groups will be calculated after testing

CONTACTS AND LOCATIONS:
Overall Officials: Thi Huyen Thuong Dang, Principal Investigator — Ho Chi Minh University Medical Center; Ngoc Tai Tran, Doctor, Study Director — Ho Chi Minh University Medical Center
Locations (1):
- Ho Chi Minh University Medical Center, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided
We will share study protocol, SAP, ICF, CSR